CLINICAL TRIAL: NCT02576509
Title: A Randomized, Multi-center Phase III Study of Nivolumab Versus Sorafenib as First-Line Treatment in Patients With Advanced Hepatocellular Carcinoma (CheckMate 459: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 459)
Brief Title: An Investigational Immuno-therapy Study of Nivolumab Compared to Sorafenib as a First Treatment in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-459
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental): Nivolumab specified dose on specified days
  Interventions: Drug: Nivolumab
- Sorafenib (Active Comparator): Sorafenib specified dose on specified days
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Nivolumab — Specified Dose on Specified Days
  Arms: Nivolumab
Drug: Sorafenib — Specified Dose on Specified Days
  Arms: Sorafenib

SUMMARY:
The purpose of this study is to determine if nivolumab or sorafenib is more effective in the treatment of Advanced Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced hepatocellular carcinoma, not eligible for surgical and/or locoregional therapies; or progressive disease after surgical and /or locoregional therapies
* Locoregional therapy for hepatocellular carcinoma (HCC) must be completed at least 4 weeks prior to the baseline scan
* Child-Pugh Class A
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Prior liver transplant
* Active, known, or suspected autoimmune disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (138):
- United States (17):
  - Local Institution - 0066, Birmingham, Alabama
  - Local Institution - 0020, Los Angeles, California
  - Local Institution - 0015, San Francisco, California
  - Local Institution - 0084, San Francisco, California
  - Local Institution - 0061, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Local Institution - 0083, New York, New York
  - Local Institution - 0093, New York, New York
  - Local Institution - 0016, Charlotte, North Carolina
  - Local Institution - 0095, Philadelphia, Pennsylvania
  - Local Institution - 0019, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Local Institution - 0017, San Antonio, Texas
  - Scott & White Memorial Hospital And Clinic, Temple, Texas
  - Local Institution - 0026, Seattle, Washington
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - Local Institution - 0050, Madison, Wisconsin
- Australia (6):
  - Local Institution - 0005, Camperdown, New South Wales
  - Local Institution - 0007, Adelaide, South Australia
  - Local Institution - 0001, Clayton, Victoria
  - Local Institution - 0002, Heidelberg, Victoria
  - Local Institution - 0003, Prahran, Victoria
  - Local Institution - 0008, Nedlands, Western Australia
- Austria (2):
  - Local Institution - 0039, Graz
  - Local Institution - 0038, Vienna
- Belgium (3):
  - Local Institution - 0075, Brussels
  - Local Institution - 0091, Leuven
  - Local Institution - 0077, Liège
- Canada (3):
  - Local Institution - 0043, Calgary, Alberta
  - Local Institution - 0044, Vancouver, British Columbia
  - Local Institution - 0042, Québec, Quebec
- China (24):
  - Local Institution - 0164, Hefei, Anhui
  - Local Institution - 0139, Beijing, Beijing Municipality
  - Local Institution - 0137, Beijing, Beijing Municipality
  - Local Institution - 0140, Beijing, Beijing Municipality
  - Local Institution - 0141, Beijing, Beijing Municipality
  - Local Institution - 0152, Fuzhou, Fujian
  - Local Institution - 0161, Guangzhou, Guangdong
  - Local Institution - 0157, Guangzhou, Guangdong
  - Local Institution - 0144, Guangzhou, Guangdong
  - Local Institution - 0158, Nanning, Guangxi
  - Local Institution - 0142, Harbin, Heilongjiang
  - Local Institution - 0148, Changsha, Hunan
  - Local Institution - 0162, Changsha, Hunan
  - Local Institution - 0169, Changzhou, Jiangsu
  - Local Institution - 0135, Nanjing, Jiangsu
  - Local Institution - 0136, Changchun, Jilin
  - Local Institution - 0163, Changchun, Jilin
  - Local Institution - 0166, Dalian, Liaoning
  - Local Institution - 0138, Xi'an, Shan3xi
  - Local Institution - 0145, Shanghai, Shanghai Municipality
  - Local Institution - 0151, Shanghai, Shanghai Municipality
  - Local Institution - 0159, Tianjin, Tianjin Municipality
  - Local Institution - 0173, Hangzhou, Zhejiang
  - Local Institution - 0146, Hangzhou, Zhejiang
- Czechia (3):
  - Local Institution - 0029, Brno
  - Local Institution - 0027, Hradec Králové
  - Local Institution - 0028, Olomouc
- France (8):
  - Local Institution - 0071, La Tronche
  - Local Institution - 0072, Lille
  - Local Institution - 0069, Lyon
  - Local Institution - 0073, Montpellier
  - Local Institution - 0067, Paris
  - Local Institution - 0068, Pessac
  - Local Institution - 0070, Rennes
  - Local Institution - 0074, Toulouse
- Germany (9):
  - Local Institution - 0036, Berlin
  - Local Institution - 0037, Essen
  - Local Institution - 0167, Frankfurt
  - Local Institution - 0034, Hamburg
  - Local Institution - 0031, Leipzig
  - Local Institution - 0035, Mainz
  - Local Institution - 0033, Munich
  - Local Institution - 0032, Regensburg
  - Local Institution - 0030, Tübingen
- Hong Kong (2):
  - Local Institution - 0011, Hong Kong
  - Local Institution - 0012, Hong Kong
- Israel (4):
  - Local Institution - 0082, Haifa
  - Local Institution - 0060, Jerusalem
  - Local Institution - 0058, Petah Tikva
  - Local Institution - 0059, Tel Aviv
- Italy (5):
  - Local Institution - 0054, Benevento
  - Local Institution - 0062, Bergamo
  - Local Institution - 0055, Milan
  - Local Institution - 0063, Orbassano
  - Local Institution - 0064, Siena
- Japan (19):
  - Local Institution - 0100, Chiba, Chiba
  - Local Institution - 0103, Matsuyama, Ehime
  - Local Institution - 0107, Kurume-shi, Fukuoka
  - Local Institution - 0127, Ogaki-shi, Gifu
  - Local Institution - 0102, Sapporo, Hokkaido
  - Local Institution - 0130, Sapporo, Hokkaido
  - Local Institution - 0105, Kanazawa, Ishikawa-ken
  - Local Institution - 0110, Kawasaki-shi, Kanagawa
  - Local Institution - 0112, Yokohama, Kanagawa
  - Local Institution - 0104, Yokohama, Kanagawa
  - Local Institution - 0111, Kyoto, Kyoto
  - Local Institution - 0106, Osaka-Sayama-Shi, Osaka
  - Local Institution - 0113, Suita, Osaka
  - Local Institution - 0115, Saga, Saga-ken
  - Local Institution - 0131, Chiyoda-ku, Tokyo
  - Local Institution - 0114, Mitaka-shi, Tokyo
  - Local Institution - 0108, Musashino-shi, Tokyo
  - Local Institution - 0126, Shinjuku-ku, Tokyo
  - Local Institution - 0101, Hiroshima
- Poland (3):
  - Local Institution - 0023, Gdansk
  - Local Institution - 0056, Warsaw
  - Local Institution - 0045, Wroclaw
- Local Institution - 0096, Moscow, Russia
- Singapore (2):
  - Local Institution - 0013, Singapore
  - Local Institution - 0014, Singapore
- South Korea (8):
  - Local Institution - 0117, Seoul, Seocho-gu
  - Local Institution - 0125, Daegu
  - Local Institution - 0116, Goyang-si
  - Local Institution - 0118, Jeollanam-do
  - Local Institution - 0123, Seoul
  - Local Institution - 0119, Seoul
  - Local Institution - 0122, Seoul
  - Local Institution - 0124, Seoul
- Spain (4):
  - Local Institution - 0065, Alicante
  - Local Institution - 0085, Majadahonda - Madrid
  - Local Institution - 0009, Pamplona
  - Local Institution - 0010, Santiago Compostela
- Sweden (2):
  - Local Institution - 0088, Gothenburg
  - Local Institution - 0087, Stockholm
- Switzerland (2):
  - Local Institution - 0040, Basel
  - Local Institution - 0041, Bern
- Taiwan (7):
  - Local Institution - 0129, Kaohsiung County
  - Local Institution - 0133, Taichung
  - Local Institution - 0121, Tainan
  - Local Institution - 0132, Tainan
  - Local Institution - 0099, Taipei
  - Local Institution - 0120, Taipei
  - Local Institution - 0128, Taoyuan
- United Kingdom (4):
  - Local Institution - 0080, London, Greater London
  - Local Institution - 0078, London, Greater London
  - Local Institution - 0079, Glasgow, Lanarkshire
  - Local Institution - 0081, Liverpool

REFERENCES:
- [Derived] Zhou X, Cao J, Topatana W, Xie T, Chen T, Hu J, Li S, Juengpanic S, Lu Z, Zhang B, Wang K, Feng X, Shen J, Chen M. Evaluation of PD-L1 as a biomarker for immunotherapy for hepatocellular carcinoma: systematic review and meta-analysis. Immunotherapy. 2023 Apr;15(5):353-365. doi: 10.2217/imt-2022-0168. Epub 2023 Feb 27. PMID 36852452
- [Derived] Li Y, Liang X, Li H, Chen X. Atezolizumab plus bevacizumab versus nivolumab as first-line treatment for advanced or unresectable hepatocellular carcinoma: A cost-effectiveness analysis. Cancer. 2022 Nov 15;128(22):3995-4003. doi: 10.1002/cncr.34457. Epub 2022 Sep 16. PMID 36111952
- [Derived] Shi J, Liu J, Tu X, Li B, Tong Z, Wang T, Zheng Y, Shi H, Zeng X, Chen W, Yin W, Fang W. Single-cell immune signature for detecting early-stage HCC and early assessing anti-PD-1 immunotherapy efficacy. J Immunother Cancer. 2022 Jan;10(1):e003133. doi: 10.1136/jitc-2021-003133. PMID 35101942
- [Derived] Yau T, Park JW, Finn RS, Cheng AL, Mathurin P, Edeline J, Kudo M, Harding JJ, Merle P, Rosmorduc O, Wyrwicz L, Schott E, Choo SP, Kelley RK, Sieghart W, Assenat E, Zaucha R, Furuse J, Abou-Alfa GK, El-Khoueiry AB, Melero I, Begic D, Chen G, Neely J, Wisniewski T, Tschaika M, Sangro B. Nivolumab versus sorafenib in advanced hepatocellular carcinoma (CheckMate 459): a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2022 Jan;23(1):77-90. doi: 10.1016/S1470-2045(21)00604-5. Epub 2021 Dec 13. PMID 34914889
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab 240 mg: Nivolumab 240 mg intravenously (IV) every 2 weeks until disease progression or unacceptable toxicity
- Sorafenib 400 mg: Sorafenib 400 mg orally (PO) twice a day (BID) until disease progression or unacceptable toxicity
Period: Pre-Treatment Period
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Started (Started = Assigned to treatment (randomized/enrolled)) | 371 | 372
Completed (Completed = Entering treatment period) | 367 | 363
Not Completed | 4 | 9
Not completed — Participant request to stop therapy | 0 | 2
Not completed — Participant withdrew consent | 1 | 5
Not completed — Participant no longer meets criteria | 3 | 2
Period: Treatment Period
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Started (Started = Received treatment) | 367 | 363
Completed | 0 | 0
Not Completed | 367 | 363
Not completed — Disease progression | 263 | 244
Not completed — Study drug toxicity | 37 | 41
Not completed — Death | 1 | 1
Not completed — Adverse event unrelated to study drug | 39 | 41
Not completed — Participant request to stop treatment | 8 | 18
Not completed — Participant withdrew consent | 3 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Maximum clinical benefit | 1 | 0
Not completed — Poor/non-compliance | 1 | 1
Not completed — Participant no longer meets criteria | 1 | 0
Not completed — Other reason | 12 | 8
Not completed — NOT REPORTED | 1 | 0
Not completed — Administrative reason by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg | Total
Number analyzed (Participants) | 371 | 372 | 743
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 185 | 176 | 361
  >=65 years | 186 | 196 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (10.61) | 64.5 (10.91) | 64.2 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 314 | 317 | 631
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 15
  Not Hispanic or Latino | 180 | 170 | 350
  Unknown or Not Reported | 186 | 192 | 378
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 165 | 167 | 332
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 199 | 196 | 395
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death due to any cause in all randomized participants. Participants who are alive will be censored at the last known alive dates.
  Based on Kaplan-Meier Estimates.
Time Frame: time from the date of randomization to the date of death due to any cause, assessed up to June 2019 (approximately 41 months)
Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Number analyzed (Participants) | 371 | 372
Months | 16.39 [13.93 to 18.37] | 14.69 [11.89 to 17.22]
Statistical Analysis 1: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Superiority; p = 0.0752, Log Rank — A priori threshold for statistical significance is 0.0419; Log-rank Test stratified by the stratification factors as entered into the IVRS; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.71 to 1.02] — Nivolumab over Sorafenib; Stratified Cox proportional hazard model; 95.81% CI ADJUSTED FOR MULTIPLICITY: (0.72 to 1.02)

2. Secondary Outcome: Objective Response Rate (ORR) Per BICR RECIST 1.1
Description: ORR is defined as the proportion of participants whose best overall response (BOR) is either a complete response (CR) or partial response (PR). BOR is defined as the best response designation, as determined based on BICR-assessed tumor response according to RECIST 1.1, recorded between the date of randomization and the date of first objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. For participants without documented progression or subsequent anti-cancer therapy, all available response designations will contribute to the BOR determination. For a BOR of CR or PR, the initial response assessment must be confirmed by a consecutive assessment no less than 4 weeks (28 days) later.
  Estimate of (Nivolumab - Sorafenib) is based on CMH method of weighting, stratified by stratification factors
Time Frame: the date of randomization and the date of first objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first, assessed up to May 2019 (approximately 40 months)
Population: all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Number analyzed (Participants) | 371 | 372
Percentage of participants | 15.4 [11.8 to 19.4] | 7.0 [4.6 to 10.1]
Statistical Analysis 1: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — no test was performed due to OS p-value result above the prior threshold; Difference of ORRs = 8.3, 95% CI 2-sided [3.9 to 12.7] — Estimate of (Nivolumab - Sorafenib) is based on CMH method of weighting, stratified by stratification factors
Statistical Analysis 2: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — no test was performed due to OS p-value result above the prior threshold; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.48 to 3.92] — Nivolumab over Sorafenib; Mantel-Haenszel estimator

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression as assessed by BICR according to RECIST 1.1 or death due to any cause in all randomized participants. Participants who die without a reported prior progression and without initiation of subsequent anti-cancer therapy will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last tumor assessment. Participants who did not have baseline tumor assessment will be censored on the date they were randomized. Participants who did not have any on study tumor assessments and did not die will be censored on the date they were randomized. Participants who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last tumor assessment prior to subsequent anti-cancer therapy.
Time Frame: time from the date of randomization to the date of the first objectively documented tumor progression or death, assessed up to May 2019 (approximately 40 months)
Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Number analyzed (Participants) | 371 | 372
Months | 3.68 [3.06 to 3.88] | 3.75 [3.71 to 4.47]
Statistical Analysis 1: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — no test was performed due to OS p-value result above the prior threshold; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.79 to 1.10] — Nivolumab over Sorafenib; Stratified Cox proportional hazard model

4. Secondary Outcome: Efficacy Based on PD-L1 Expression - OS and PFS
Description: PD-L1 expression is defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per Dako PD-L1 IHC assay unless otherwise specified. This is referred as quantifiable PD-L1 expression. If the PD-L1 staining could not be quantified, it is further classifies as:
  Indeterminate: Tumor cell membrane staining hampered for reasons attributed to the biology of the tumor biopsy specimen and not because of improper sample preparation or handling.
  Not evaluable: Tumor biopsy specimen was not optimally collected or prepared (e.g. PD-L1 expression is neither quantifiable nor indeterminate).
  PD-L1 status is a dichotomized variable using an X% cut-off for quantifiable PD-L1 expression:
  * PD-L1 > X %: ≥ X % PD-L1 expression
  * PD-L1 < X %: < X % PD-L1 expression where X% denotes the PD-L1 expression cut-off of 1%. Additional cut off values may also be explored.
  Confidence interval based on the Clopper and Pearson method.
Time Frame: as for outcome 2
Population: all randomized participants with a >=1% PD-L1 expression all randomized participants with a <1% PD-L1 expression all randomized participants without PD-L1 quantifiable
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Number analyzed (Participants) | 371 | 372
Months
  >=1%, OS: number analyzed (Participants) | 71 | 64
  >=1%, OS | 16.07 [8.41 to 22.34] | 8.62 [5.72 to 16.30]
  >=1%, PFS: number analyzed (Participants) | 71 | 64
  >=1%, PFS | 3.84 [2.10 to 7.62] | 3.58 [1.97 to 5.36]
  <1%, OS: number analyzed (Participants) | 295 | 300
  <1%, OS | 16.72 [13.93 to 18.56] | 15.24 [12.58 to 18.10]
  <1%, PFS: number analyzed (Participants) | 295 | 300
  <1%, PFS | 3.61 [2.43 to 3.81] | 3.75 [3.71 to 5.32]
  without PD-L1 quantifiable, OS: number analyzed (Participants) | 5 | 8
  without PD-L1 quantifiable, OS | 16.23 [5.82 to NA] — Upper limit cannot be estimated based on the data | 22.05 [1.77 to NA] — Upper limit cannot be estimated based on the data
  without PD-L1 quantifiable, PFS: number analyzed (Participants) | 5 | 8
  without PD-L1 quantifiable, PFS | 2.00 [1.87 to NA] — Upper limit cannot be estimated based on the data | 6.13 [1.08 to 11.17]
Statistical Analysis 1: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — PD-L1 >= 1%, OS; no test was performed; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.54 to 1.19] — Nivolumab over Sorafenib
Statistical Analysis 2: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — PD-L1 >=1%, PFS; no test was performed; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.48 to 1.03] — Nivolumab over Sorafenib
Statistical Analysis 3: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — PD-L1 <1%, OS; no test was performed; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.02] — Nivolumab over Sorafenib
Statistical Analysis 4: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — PD-L1 <1%, PFS; no test was performed; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.81 to 1.17] — Nivolumab over Sorafenib
Statistical Analysis 5: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — without PD-L1 quantifiable, OS; no test was performed; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.34 to 4.74] — Nivolumab over Sorafenib
Statistical Analysis 6: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — without PD-L1 quantifiable, PFS; no test was performed; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.27 to 3.52] — Nivolumab over Sorafenib

5. Secondary Outcome: Efficacy Based on PD-L1 Expression - ORR
Description: as for outcome 4
Time Frame: as for outcome 2
Population: all randomized participants with a >=1% PD-L1 expression all randomized participants with a <1% PD-L1 expression all randomized participants without PD-L1 quantifiable Note: odds ratio for participants without PD-L1 quantifiable cannot be estimated based on the data
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
Number analyzed (Participants) | 371 | 372
Percentage of participants
  >=1%, ORR: number analyzed (Participants) | 71 | 64
  >=1%, ORR | 28.2 [18.1 to 40.1] | 9.4 [3.5 to 19.3]
  <1%, ORR: number analyzed (Participants) | 295 | 300
  <1%, ORR | 12.2 [8.7 to 16.5] | 6.7 [4.1 to 10.1]
  without PD-L1 quantifiable, ORR: number analyzed (Participants) | 5 | 8
  without PD-L1 quantifiable, ORR | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 36.9]
Statistical Analysis 1: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — PD-L1 >=1%, ORR; no test was performed; Odds Ratio (OR) = 3.79, 95% CI 2-sided [1.41 to 10.17] — Odds ratio (Nivolumab over Sorafenib) and associated unstratified 95% exact CI
Statistical Analysis 2: Comparison: Nivolumab 240 mg vs Sorafenib 400 mg; Test type: Other — PD-L1 <1%, ORR; no test was performed; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.10 to 3.45] — Odds ratio (Nivolumab over Sorafenib) and associated unstratified 95% exact CI

ADVERSE EVENTS:
Time Frame: All cause mortality was collected from randomization up to last survival follow up (approximately up to 98 months). Serious and non-serious adverse events were collected from first dose till 100 days after last dose of study therapy (up to approximately 95 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Nivolumab 240 mg | Sorafenib 400 mg
All-Cause Mortality (participants affected / at risk) | 321/371 | 335/372
Serious Adverse Events (participants affected / at risk) | 216/367 | 216/363
Other Adverse Events (participants affected / at risk) | 339/367 | 351/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 240 mg (N=367) | Sorafenib 400 mg (N=363)
Anaemia (Blood and lymphatic system disorders) | 8 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Eyelid function disorder (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 11
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 9 | 7
Colitis (Gastrointestinal disorders) | 5 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 0
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 6
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 8
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 6
Varices oesophageal (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Asthenia (General disorders) | 0 | 3
Catheter site related reaction (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 4
General physical health deterioration (General disorders) | 8 | 14
Hypothermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 7
Sudden death (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 1 | 1
Biloma (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 4 | 4
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 10 | 7
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 3
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 3 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 3 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Genitourinary tract infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 4
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 2
Septic shock (Infections and infestations) | 0 | 2
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Viral pharyngitis (Infections and infestations) | 1 | 0
Virologic failure (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 3 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 2 | 0
Occult blood positive (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 69 | 70
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 3 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Cognitive disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 4
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 6 | 6
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Malignant spinal cord compression (Nervous system disorders) | 1 | 0
Middle cerebral artery stroke (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 5
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Agonal respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Assisted suicide (Surgical and medical procedures) | 0 | 1
Aneurysm ruptured (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 240 mg (N=367) | Sorafenib 400 mg (N=363)
Anaemia (Blood and lymphatic system disorders) | 35 | 30
Hypothyroidism (Endocrine disorders) | 29 | 12
Abdominal distension (Gastrointestinal disorders) | 15 | 22
Abdominal pain (Gastrointestinal disorders) | 69 | 82
Abdominal pain upper (Gastrointestinal disorders) | 42 | 50
Ascites (Gastrointestinal disorders) | 46 | 44
Constipation (Gastrointestinal disorders) | 50 | 52
Diarrhoea (Gastrointestinal disorders) | 100 | 191
Nausea (Gastrointestinal disorders) | 62 | 70
Stomatitis (Gastrointestinal disorders) | 16 | 25
Vomiting (Gastrointestinal disorders) | 36 | 40
Asthenia (General disorders) | 40 | 43
Fatigue (General disorders) | 103 | 117
Oedema peripheral (General disorders) | 43 | 41
Pyrexia (General disorders) | 71 | 58
Nasopharyngitis (Infections and infestations) | 33 | 23
Upper respiratory tract infection (Infections and infestations) | 29 | 15
Alanine aminotransferase increased (Investigations) | 51 | 38
Amylase increased (Investigations) | 26 | 14
Aspartate aminotransferase increased (Investigations) | 84 | 60
Blood alkaline phosphatase increased (Investigations) | 19 | 17
Blood bilirubin increased (Investigations) | 41 | 48
Lipase increased (Investigations) | 38 | 27
Platelet count decreased (Investigations) | 17 | 28
Weight decreased (Investigations) | 34 | 68
Decreased appetite (Metabolism and nutrition disorders) | 77 | 135
Hyperglycaemia (Metabolism and nutrition disorders) | 21 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 | 31
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 12
Dizziness (Nervous system disorders) | 23 | 14
Headache (Nervous system disorders) | 24 | 33
Insomnia (Psychiatric disorders) | 32 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 47
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 71
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 21
Erythema (Skin and subcutaneous tissue disorders) | 5 | 31
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 29 | 181
Pruritus (Skin and subcutaneous tissue disorders) | 88 | 51
Rash (Skin and subcutaneous tissue disorders) | 75 | 59
Hypertension (Vascular disorders) | 33 | 85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02576509/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT02576509/SAP_002.pdf